CLINICAL TRIAL: NCT07313241
Title: Phase II Trial of PSA Response-based Androgen Deprivation Therapy and Nodal Coverage for Prostate Cancer Early Salvage Radiotherapy (RANGER)
Acronym: (RANGER)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Aurelie Garant, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20251220
Record Dates: First submitted 2025-12-16; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm: PSA Response Adapted Salvage Radiotherapy (Experimental): All participants initially receive prostate fossa radiotherapy (RT) using stereotactic ultra-hypofractionated dosing (32.5 Gy in 5 fractions over 2-4 weeks) delivered via the Ethos™ online adaptive platform.
  At approximately 5 weeks post-RT initiation, PSA response is assessed:
  * Responders: Patients with PSA <0.05 ng/mL or a decrease of ≥0.2 ng/mL compared to pre-RT PSA will undergo observation without further immediate therapy.
  * Non-Responders: Patients not meeting response criteria will receive sequential pelvic nodal RT (25 Gy in 5 fractions over ≤4 weeks) plus androgen deprivation therapy (ADT) for 4 months. Pelvic nodal RT begins within 14 days after response assessment. ADT (GnRH agonists/antagonists, e.g., leuprolide, goserelin, degarelix) will be started before or within 14 days of pelvic nodal RT initiation.
  Interventions: Radiation: Prostate Fossa Radiotherapy; Radiation: Pelvic nodal Radiotherapy; Drug: Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Radiation: Prostate Fossa Radiotherapy — Stereotactic ultra hypofractionanted radiotherapy delivered to the prostate fossa using the Ethos online adaptive platform. Total dose of 32.5 Gy administered in 5 fractions over 2-4 weeks.
Radiation: Pelvic nodal Radiotherapy — Sequential pelvic nodal radiotherapy delivered only to PSA non responders. Dose of 25 Gy given in 5 fractions over 4 weeks using the same stereotactic technique as prostate fossa RT.
Drug: Androgen Deprivation Therapy (ADT) — GnRH agonist or antagonist (leuprolide, goserelin, degarelix) administered as per institutional standard. Therapy duration is 4 months, starting before or within 14 days of pelvic nodal RT initiation.

SUMMARY:
This Phase II, single arm study evaluates a PSA-response-adapted approach to salvage radiotherapy after radical prostatectomy for prostate cancer. All participants will receive hypo-fractionated stereotactic radiotherapy to the prostate fossa. At 5 weeks, biochemical response will be assessed. responders will proceed to observation, while non responders will receive sequential pelvic nodal radiotherapy and 4 months of androgen deprivation therapy (ADT). The study aims to determine whether this response base approach achieves non inferior 2 year freedom from progression compared with historical outcomes using routine pelvic nodal radiotherapy and ADT in all patients.

DETAILED DESCRIPTION:
After radical prostatectomy, many men experience biochemical recurrence despite having no visible metastatic disease. Standard salvage radiotherapy is effective but often includes universal use of androgen deprivation therapy and pelvic nodal radiotherapy, which may expose many patients to unnecessary toxicity.

The study evaluates a response adapted strategy using hypo fractionated or ultra hypo fractionated prostate fossa radiotherapy delivered on the Ethos adaptive radiotherapy platform. All participants will undergo 5 fractions of prostate fossa radiotherapy. At 5 weeks from treatment initiation, biochemical response will be defined as PSA <0.05 ng/mL or a 0.2 ng/mL decrease from pre-treatment PSA. Responders will undergo observation. Non responders will receive sequential pelvic nodal stereotactic radiotherapy in 5 fractions and a 4 month course of ADT.

Primary objective is to determine whether PSAA response adapted escalation achieves non inferior 2 year freedom from progression compared with historical control data. Secondary outcomes include patient reported hormonal, urinary, and bowel symptoms (EPIC-26), as well as physician graded gastrointestinal and genitourinary toxicities. Exploratory objectives include evaluating locoregional and distant failure.

This approach may reduce unnecessary toxicity for responders whole allowing early selective intensification for non responders, shortening total treatment duration for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥18 years with histologically confirmed prostate adenocarcinoma treated with prostatectomy in the localized setting within 10 years, with post-operative PSA (persistent or rising) of ≥0.05ng/mL.
* Radical prostatectomy ≥4 months prior to enrollment without nodal involvement (pN0 or pNx)
* Performance status ECOG 0-2
* No definite evidence of regional or distant metastatic disease by at least pelvic imaging within 90 days of registration. Equivocal findings are allowed at investigator discretion. Imaging is specified as follows:

  * PSA>=0.2ng/mL: positron emission tomography (PET) with FDA-approved advanced imaging agent for prostate cancer (e.g. PSMA) required.
  * PSA <0.2 n/gm: PET with above noted agents OR conventional CT or MRI at investigator discretion.
* All sexually active men must agree to use adequate contraception for the duration of study therapies and a period of 60 days thereafter. Should a female partner of a trial participant become pregnant or suspect she is pregnant while the subject is participating in this study, the patient should inform his treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior androgen deprivation therapy (ADT) > 3 months OR anti-androgen therapy (AAT) of > 30 days. For shorter courses of either, at least 30 day "wash out" period is required with confirmation of resolved castration of testosterone to >50ng/mL.
* Ongoing testosterone replacement therapy (TRT) with refusal to discontinue (must be stopped with demonstration of detectable PSA ≥0.05ng/mL and non-castrate testosterone >50ng/mL after 14 days of TRT cessation)
* Prior pelvic radiotherapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* History of bladder neck or urethral stricture requiring procedural intervention.
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to actively interfere with the safety or efficacy assessments of this study in the investigator's view.
* Active inflammatory bowel disease requiring recurring systemic or steroid/enema therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only study- Prostate cancer with rising PSA after surgical removal of the prostate and without evidence of disease beyond the prostate bed
Enrollment: 68 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2030-11-14 (Estimated); Study Completion 2030-11-14 (Estimated)

PRIMARY OUTCOMES:
Freedom from failure | 2 years from end of radiotherapy
  first occurrence of rise of PSA of 2 ng/dL above post-salvage RT nadir, clinical progression (local/regional/distant) or death due to any cause.

SECONDARY OUTCOMES:
EPIC-26 hormonal summary domain score | Baseline and regular intervals during 2 year follow up
  Patient reported hormonal symptom severity measure by the EPIC-26 questionnaire
EPIC-26 Genitourinary (GU) summary domain score | Baseline and regular intervals during 2 year follow up
  Patient reported genitourinary symptom severity measure by EPIC-26
EPIC-26 Gastrointestinal (GI) summary domain score | Baseline and regular intervals during 2 year follow up
  Patient reported gastrointestinal severity measured by EPIC-26
CTCAE v5.0 toxicity GU and GI | Baseline and regular intervals during 2 year follow up
  GI and GU adverse events will be assessed and graded according to the National Cancer Institute Common Technology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Aurelie Garant, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center-Dallas, Dallas, Texas, United States